CLINICAL TRIAL: NCT07079683
Title: A Randomized Clinical Trial to Determine the Effect of a Toothpaste Containing Enzymes Blend of Alpha-Amylase and Gluco-Amylase on Dental Biofilm Plaque Accumulation in Healthy Adults Over a 28-Day Period of Product Use
Brief Title: RCT: Enzyme Blend Toothpaste on Dental Biofilm Plaque Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NZ-2022-04
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Dental Biofilm Accumulation
Keywords: RCT; Toothpaste; Enzymes; Biofilm

STUDY DESIGN:
Intervention Model Description: This will be a single center, placebo controlled, double-blind, randomized, two-treatment arm, parallel design, clinical study. Study subjects will be aged 18 years or older, non-smokers, in good general health with generalized mild to moderate plaque-induced gingivitis and ≥ 20 natural teeth. The use of a Washout period prior to Baseline will be included in this design so that subjects avoid use of antimicrobial mouth rinses, dentifrices or other dental products that might affect a subject's plaque or gingivitis status. Subjects will be asked to use a marketed fluoride-free toothpaste and soft bristle toothbrush as their only oral hygiene regimen. A minimum of 7 days lead-in period is appropriate to allow subjects to comply with study and lifestyle restrictions prior to Baseline Visit. Subjects must meet all study criteria at both the Screening and Baseline visits to be eligible for participation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Lab personnel were also blinded when analyzing exploratory markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo toothpaste without enzymes (Placebo Comparator): Placebo toothpaste without enzymes to be used twice a day, morning and evening, (one minute) at a dose of approximately 1.5 g/toothbrushing (full ribbon of toothpaste) for the 28-day study duration.
  Interventions: Other: Toothpaste Product
- BioFresh Clean toothpaste containing a blend of alpha-amylase and gluco-amylase enzymes (Experimental): BioFresh toothpaste containing a blend of alpha-amylase and gluco-amylase enzymes to be used twice a day, morning and evening, (one minute) at a dose of approximately 1.5 g/toothbrushing (full ribbon of toothpaste) for the 28-day study duration.
  Interventions: Other: Toothpaste Product

INTERVENTIONS:
Other: Toothpaste Product — BioFresh toothpaste containing a blend of alpha-amylase and gluco-amylase enzymes to be used twice a day, morning and evening, (one minute) at a dose of approximately 1.5 g/toothbrushing (full ribbon of toothpaste) for the 28-day study duration.
  Arms: BioFresh Clean toothpaste containing a blend of alpha-amylase and gluco-amylase enzymes
Other: Toothpaste Product — Placebo toothpaste containing no enzymes to be used twice a day, morning and evening, (one minute) at a dose of approximately 1.5 g/toothbrushing (full ribbon of toothpaste) for the 28-day study duration.
  Arms: Placebo toothpaste without enzymes

SUMMARY:
The aim of the study is to investigate whether brushing twice a day with a toothpaste (Biofresh Clean) containing a blend of alpha-amylase and gluco-amylase improves oral health outcomes over a 14-day period.

The primary objective is to evaluate if the enzyme-containing toothpaste has an effect on dental plaque accumulation compared to placebo following 28 days of use.

The secondary objectives are to:

* Evaluate if the enzyme-containing toothpaste has an effect on dental plaque accumulation compared to placebo at Days 1 and 14
* Evaluate if the enzyme-containing toothpaste has an effect on gumline and proximal plaque severity compared to placebo at Days 1, 14 and 28
* Evaluate if the enzyme-containing toothpaste has an effect on whole mouth Gingivitis as well as gumline and proximal Gingivitis severity compared to placebo at Days 14 and 28

The exploratory variables are to investigate if the enzyme-containing toothpaste results in:

* Shift in detected oral bacterial species of interest at Screening and Baseline to Days 14 and 28, based on microbial DNA-extraction and microbial whole genome sequencing compared to placebo.
* Shift in immune markers (IL-1β, , IL-8 and MIF) at Screening and Baseline to Days 14 and 28, based on electrochemiluminescence assay compared to placebo.
* Difference in performance attributes compared to placebo based on End of Study Post-product use questionnaire after 28 days of product use.

The safety objective is to investigate safety and tolerability of brushing twice daily based on treatment emergent adverse events.

Target Population Randomized subjects are generally healthy males and females (18-65y) with at least 20 natural teeth, A gingival index score of ≥ 1.0, according to the Löe-Silness Gingival Index at baseline and a plaque index score ≥ 1.95 according to the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index..

Researchers will compare Biofresh Clean Toothpaste to an identically packaged and labelled placebo to see if Biofresh Clean Toothpaste reduces dental plaque accumulation and Gingivitis.

Participants will:

* Brush teeth for one minute twice per day (morning and evening) with either 1.5g of Biofresh Clean toothpaste or identical placebo toothpaste over 14-days.
* Visit the dental clinic on 5 occasions: 1. Screening visit to assess eligibility; 2. Baseline visit; 3. Day 1 Visit; 4. Day 14 visit; 5. Day 28 visit

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy males and females 18-65 years of age.
2. Able to read, sign and receive a copy of the signed informed consent form.
3. Willing and able to comply with scheduled visits, treatment plan and other study procedures.
4. Subject is in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the subject's safety, wellbeing or the outcome of the study.
5. At the Screening Visit (Visit 1):

   1. Have at least 20 natural teeth with scorable facial and lingual surfaces. (A scorable surface is defined as having 2/3rds of the natural tooth surface gradable for the selected clinical indices. The following should not be included in the evaluable surface count- third molars; fully crowned/extensively restored, grossly carious, orthodontically banded/bonded or abutment teeth; surfaces with calculus deposits which, in the opinion of the clinical examiner, would interfere with the baseline assessments of the selected clinical indices.)
   2. Subject with generalized mild-moderate plaque-induced gingivitis, in the opinion of the clinical examiner, as confirmed by visual examinations.
6. At Screening Visit (Visit 1):

   1. A gingival index score of ≥ 1.0, according to the Löe-Silness Gingival Index.
   2. A plaque index score ≥ 1.95 according to the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index, following 8 to 16 hours plaque accumulation period.
7. Willing to refrain from all oral hygiene 8-16 hours prior to each study visit, refrain from eating within 4 hours prior to each study visit and discontinue drinking 30 minutes prior to each study visit.
8. Willing to refrain from using chewing gum, breath mints and lozenges for the duration of the study.
9. Willing to refrain from the use of chemotherapeutic antiplaque/antigingivitis products containing antibacterial agents such as, but not limited to, amine fluoride, chlorhexidine, stannous fluoride, essential oils, cetylpyridinium chloride, etc. and other oral hygiene products during the study.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Have any medical condition that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.
2. History of allergy or significant adverse events following use of oral hygiene products such as toothpastes, mouth rinses, breath mints, lozenges, or chewing gum or their ingredients.
3. A subject who is pregnant or intending to become pregnant over the duration of the study (self-reported).
4. A subject who is breastfeeding.
5. Self-reported serious medical conditions.
6. Uncontrolled diabetes or hypertension.
7. Antibiotic or anti-inflammatory medication within 30 days of screening visit. 8. Smokers or users of other nicotine products.

9. Any health condition that requires prophylactic antibiotics prior to any dental procedure to prevent infective endocarditis.

10. Daily use of steroidal or non-steroidal anti-inflammatory drugs. 11. Have had antibiotic, anti-inflammatory, or chemotherapeutic antiplaque/antigingivitis therapy within 30 days of screening exams.

12. Unwilling to discontinue use of other oral hygiene products (e.g., antiplaque-antigingivitis mouthrinses or dentifrices, power toothbrushes, oral irrigators/water flossers) for the duration of the study.

13. Clinically visible active caries lesions and/or periodontitis. 14. Orthodontic appliances, including retainers, peri/oral piercings, or removable partial dentures.

15. Exhibits ≥ 30% of teeth with stage II - IV periodontitis, according to the American Academy of Periodontology revised classification system for periodontal and peri-implant diseases and conditions,8 at screening and/or baseline visit, or being actively treated for periodontal disease, and have more than three teeth with periodontal pockets depths measuring more than 5 mm. 16. Have significant intra-oral soft tissue lesions due to pathology or trauma based on a visual examination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Whole mouth dental plaque accumulation at Day 28. | Day 28
  Change in mean whole Mouth (WM) dental plaque accumulation assessed using the Lobene-Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index (PLI) with a score range from 0 to 5. A score of 0 means no plaque, while higher scores indicate increasing amounts of plaque.

SECONDARY OUTCOMES:
Whole mouth dental plaque accumulation Day 1 | Day 1
  Mean WM dental plaque accumulation is assessed using PLI with a score range from 0 to 5. A score of 0 means no plaque, while higher scores indicate increasing amounts of plaque.
Whole mouth dental plaque accumulation Day 14 | Day 14
  Mean WM dental plaque accumulation is assessed using PLI with a score range from 0 to 5. A score of 0 means no plaque, while higher scores indicate increasing amounts of plaque.
Gumline Plaque Severity Index (PSI) scores Day 1 | Day 1
  Gumline Plaque Severity Index (PSI) scores calculated from PLI scores by dividing the total number of tooth surface sites receiving scores of 3, 4 or 5 by the total number of tooth surface sites scored in the mouth. The scale is ranging from 0 to 5, with higher scores indicating a worse condition.
Gumline Plaque Severity Index (PSI) scores Day 14 | Day 14
  Gumline PSI scores calculated from PLI scores by dividing the total number of tooth surface sites receiving scores of 3, 4 or 5 by the total number of tooth surface sites scored in the mouth. The scale is ranging from 0 to 5, with higher scores indicating a worse condition.
Gumline Plaque Severity Index (PSI) scores Day 28 | Day 28
  Gumline PSI scores calculated from PLI scores by dividing the total number of tooth surface sites receiving scores of 3, 4 or 5 by the total number of tooth surface sites scored in the mouth. The scale is ranging from 0 to 5, with higher scores indicating a worse condition.
Proximal Plaque Severity Index (PSI) scores at Day 1 | Day 1
  Proximal Plaque Severity Index (PSI) scores calculated from PLI scores by dividing the total number of tooth surface sites receiving scores of 3, 4 or 5 by the total number of tooth surface sites scored in the mouth. The scale is ranging from 0 to 5, with higher scores indicating a worse condition.
Proximal Plaque Severity Index (PSI) scores Day 14 | Day 14
  Proximal PSI scores calculated from PLI scores by dividing the total number of tooth surface sites receiving scores of 3, 4 or 5 by the total number of tooth surface sites scored in the mouth. The scale is ranging from 0 to 5, with higher scores indicating a worse condition.
Proximal Plaque Severity Index (PSI) scores Day 28 | Day 28
  Proximal PSI scores calculated from PLI scores by dividing the total number of tooth surface sites receiving scores of 3, 4 or 5 by the total number of tooth surface sites scored in the mouth. The scale is ranging from 0 to 5, with higher scores indicating a worse condition.
Whole mouth Gingival Index (GI) scores Day 14 | Day 14
  Whole mouth Gingivitis Index score according to according to the Löe-Silness Gingival Index (GI) scoring it on a scale from 0 to 3, with 0 representing a healthy gingiva and 3 indicating severe inflammation.
Whole mouth Gingival Index (GI) scores Day 28 | Day 28
  Whole mouth Gingivitis Index score according to according to the Löe-Silness Gingival Index (GI) scoring it on a scale from 0 to 3, with 0 representing a healthy gingiva and 3 indicating severe inflammation.
Gumline Gingivitis Severity Index score Day 14 | Day 14
  Gumline Gingivitis Severity Index score according to the Löe-Silness Gingival Index, the proportion of tooth sites receiving the high-level GI scores of 2 and 3 at baseline will be included in the calculation to provide the Gingivitis Severity Index measures.19 Site-wise scores for whole mouth, gumline and proximal sites, will be calculated by counting the scores for the sites with baseline GI = 2 and 3 and dividing by the total number of sites assessed. The score is ranging from 0 to 3, with higher scores reflect more advanced inflammation.
Gumline Gingivitis Severity Index score Day 28 | Day 28
  Gumline Gingivitis Severity Index score according to the Löe-Silness Gingival Index, the proportion of tooth sites receiving the high-level GI scores of 2 and 3 at baseline will be included in the calculation to provide the Gingivitis Severity Index measures.19 Site-wise scores for whole mouth, gumline and proximal sites, will be calculated by counting the scores for the sites with baseline GI = 2 and 3 and dividing by the total number of sites assessed. The score is ranging from 0 to 3, with higher scores reflect more advanced inflammation.
Proximal Gingivitis Severity Index score Day 14 | Day 14
  Proximal Gingivitis Severity Index score according to the Löe-Silness Gingival Index, the proportion of tooth sites receiving the high-level GI scores of 2 and 3 at baseline will be included in the calculation to provide the Gingivitis Severity Index measures.19 Site-wise scores for whole mouth, gumline and proximal sites, will be calculated by counting the scores for the sites with baseline GI = 2 and 3 and dividing by the total number of sites assessed. The score is ranging from 0 to 3, with higher scores reflect more advanced inflammation.
Proximal Gingivitis Severity Index scores Day 28 | Day 28
  Proximal Gingivitis Severity Index score according to the Löe-Silness Gingival Index, the proportion of tooth sites receiving the high-level GI scores of 2 and 3 at baseline will be included in the calculation to provide the Gingivitis Severity Index measures.19 Site-wise scores for whole mouth, gumline and proximal sites, will be calculated by counting the scores for the sites with baseline GI = 2 and 3 and dividing by the total number of sites assessed. The score is ranging from 0 to 3, with higher scores reflect more advanced inflammation.

OTHER OUTCOMES:
Shift in bacterial species in oral microbiome | Day 14 and Day 28
  Shift in detected oral bacterial species based on microbial DNA-extraction and microbial whole genome sequencing
Shift in salivary immune markers from baseline to Day 14 and Day 28 | Day 14 and Day 28
  Shift in salivary immune markers (IL-1β, IL-8 and macrophage inhibition factor (MIF)
Product use questionnaire | 28-days
  Evaluate the effect on ....? based on a product use questionnaire (validated?) following 28 days of product use.
Safety and tolorability | 28-days
  Assess safety and tolerability of twice daily brushing based on number of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Milleman, DDS, MPA, Principal Investigator — Salus Research Inc
Locations (1):
- Salus Research Inc, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No